CLINICAL TRIAL: NCT05682222
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Dose Platform Study Investigating the Immunopharmacology of EDP1815 and EDP2939.
Brief Title: Evaluation of the Immunopharmacology of EDP1815 and EDP2939
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EDP1815-105
Record Dates: First submitted 2022-07-22; First posted 2023-01-12 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: KLH and Imiquimod Induced Skin Inflammation in Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind, placebo-controlled, platform trial to evaluate the effects of EDP1815 and EDP2939 on the systemic immune system, using intradermal KLH and topical IMQ skin challenges. A total of at least 72 healthy volunteers will be divided into 4 cohorts.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Other): EDP1815 or placebo in capsule A, dosed for 60 days. Randomization is 2:1 active:placebo.
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 2 (Other): EDP1815 or placebo in capsule B, dosed for 60 days. Randomization is 2:1 active:placebo.
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 3 (Other): EDP2939 lower dose or placebo in capsule B, dosed for 60 days. Randomization is 2:1 active:placebo.
  Interventions: Drug: EDP2939; Drug: Placebo oral capsule
- Cohort 4 (Other): EDP2939 higher dose or placebo in capsule B, dosed for 60 days. Randomization is 2:1 active:placebo.
  Interventions: Drug: EDP2939; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an essentially non-viable, non-replicating pharmaceutical preparation of a single strain of Prevotella histicola, a naturally occurring human commensal microbe.
  Arms: Cohort 1; Cohort 2
Drug: EDP2939 — EDP2939 is a pharmaceutical preparation of extracellular vesicles.
  Arms: Cohort 3; Cohort 4
Drug: Placebo oral capsule — Placebo.

SUMMARY:
A single-center, randomized, double-blind, placebo-controlled, multiple dose platform trial.

DETAILED DESCRIPTION:
This study will evaluate the pharmacodynamic effects of multiple doses of EDP1815 and EDP2939 on immunological responses to keyhole limpet hemocyanin (KLH) and imiquimod (IMQ) dermal challenges in healthy volunteers.

EDP1815 is an essentially non-live, specific strain of Prevotella histicola, a natural human commensal organism. EDP2939 is a pharmaceutical preparation of microbial extracellular vesicles.

Four cohorts of volunteers (n=18 per cohort) will be studied using different capsule formulations and doses, administered for 60 days. Volunteers will be immunised with intramuscular KLH. Intradermal KLH re-challenge and topical IMQ challenge will commence on Day 57 with serial pharmacodynamic assessments to Day 60. Responses will be evaluated using dermal imaging (laser speckled contrast imaging; LSCI, and multi-spectral photography), as well as dermal and systemic immunological biomarkers.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of giving signed informed consent, and willing to comply with requirements of the study.
* Age 18 years to 45 years, inclusive.
* Body mass index of 18 to 35 kg/m2, inclusive.
* Caucasian.
* Healthy based on medical history, physical examination, blood pressure, ECG and blood and urine laboratory tests.

Key Exclusion Criteria:

* Use of Aldara® (imiquimod cream) within 3 weeks prior to the study.
* Has previously received Immucothel® or KLH.
* Allergy to Alhydrogel® or Aldara® (imiquimod cream).
* Current or recurrent skin diseases affecting the arms or back, or extensive tattoos in these areas.
* Previous diagnosis of psoriasis.
* History of pathological scar formation (e.g. keloid scar).
* History of skin cancer (basal cell carcinoma, squamous cell carcinoma, melanoma).
* Significant bowel disease (e.g. inflammatory bowel disease, coeliac disease)
* Currently has an infection or has needed antibiotics within 6 weeks before the study.
* Current smoker of more than 5 cigarettes per day
* Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks before start of the study
* History of Schistosomiasis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
KLH-induced immune reaction. | At 24 hours after Day 57 intradermal re-challenge.
  This will be measured as basal flow (arbitrary units, AU) by LSCI.

SECONDARY OUTCOMES:
KLH-induced immune reaction - basal flow. | At 4 hours, 48 hours and 72 hours after Day 57 intradermal re-challenge.
  This will be measured as basal flow (AU) by LSCI.
KLH-induced immune reaction - flare. | At 4 hours, 24 hours, 48 hours and 72 hours after Day 57 intradermal re-challenge.
  This will be measured as flare (AU) by LSCI.
KLH-induced immune reaction - erythema. | At 4 hours, 24 hours, 48 hours and 72 hours after Day 57 intradermal re-challenge.
  This will be measured as erythema (AU) by multispectral imaging.
IMQ-induced immune reaction - basal flow. | At 24 hours, 48 hours and 72 hours after Day 57 initiation of IMQ challenge.
  This will be measured as basal flow (AU) by LSCI.
IMQ-induced immune reaction - flare. | At 24 hours, 48 hours and 72 hours after Day 57 initiation of IMQ challenge.
  This will be measured as flare (AU) by LSCI.
IMQ-induced immune reaction - erythema. | At 24 hours, 48 hours and 72 hours after Day 57 initiation of IMQ challenge.
  This will be measured as erythema (AU) by multispectral imaging.
Specific B-cell response to KLH. | After Day 57 intradermal re-challenge.
  This will be measured as anti-KLH IgM and IgG (% of baseline concentration).
Serious adverse event (SAE) and adverse event (AE) incidents. | Up to Day 74.
  SAEs and AEs assessed by: type, frequency, severity and treatment-relatedness of the event.
Number of participants with blood laboratory safety abnormalities. | Up to Day 74.
Number of participants with urinary laboratory safety abnormalities. | Up to Day 74.
Number of participants with electrocardiogram (ECG) abnormalities. | Up to Day 74.
Number of participants with vital signs abnormalities. | Up to Day 74.
Number of participants with physical examination abnormalities. | Up to Day 74.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eveleens Maarse BC, Ronner MN, Jansen MAA, Niemeyer-van der Kolk T, In 't Veld AE, Klaassen ES, Ahmad S, Itano A, McHale D, Moerland M. Immunomodulating effects of the single bacterial strain therapy EDP1815 on innate and adaptive immune challenge responses - a randomized, placebo-controlled clinical trial. Immunol Res. 2024 Aug;72(4):776-787. doi: 10.1007/s12026-024-09484-7. Epub 2024 May 15. PMID 38748319